CLINICAL TRIAL: NCT00728663
Title: Docetaxel and Cetuximab in Patients With Docetaxel-resistant Hormone-refractory Prostate Cancer (HRPC). A Multicenter Phase II Trial
Brief Title: Docetaxel and Cetuximab in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 08/07; SWS-SAKK-08-07; MERCK-SAKK-0807; SANOFI-AVENTIS-SWS-SAKK-0807; CDR0000599858
Record Dates: First submitted 2008-08-05; First posted 2008-08-06 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cetuximab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm: Cetuximab and Docetaxel (Experimental): Cetuximab: 400 mg/m2 initial dose on day 1, then 250 mg/m2 weekly starting on day 8 and Docetaxel: 75 mg/m2 day 1 of a 21 day cycle or 35 mg/m2 day 1,8,15 of a 28 day cycle
  --- for max. 24 weeks or until progression or unacceptable toxicity ---
  Interventions: Biological: cetuximab; Drug: docetaxel

INTERVENTIONS:
Biological: cetuximab — Cetuximab: 400 mg/m2 initial dose on day 1, then 250 mg/m2 weekly starting on day 8
  --- for max. 24 weeks or until progression or unacceptable toxicity ---
  Other Names: Erbitux
Drug: docetaxel — 75 mg/m2 day 1 of a 21 day cycle or 35 mg/m2 day 1,8,15 of a 28 day cycle
  --- for max. 24 weeks or until progression or unacceptable toxicity ---
  Other Names: Taxotere

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of prostate cancer by blocking blood flow to the tumor. Giving docetaxel together with cetuximab may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving docetaxel together with cetuximab and to see how well it works in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the efficacy and safety of docetaxel and cetuximab in patients with docetaxel-resistant hormone-refractory prostate cancer

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV once weekly and docetaxel IV on day 1 (3-week courses) or on days 1, 8, and 15 (4-week courses). Treatment repeats every 3 weeks for up to 8 courses or every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Metastatic adenocarcinoma of the prostate
* Must have received one of the following treatment schedules for at least 12 weeks prior to study therapy:

  * Docetaxel 75 mg/m^2 on day 1 of a 21-day course
  * Docetaxel 35 mg/m^2 on days 1, 8, and 15 of a 28-day course
* Must demonstrate hormone-resistance, defined as tumor progression after orchiectomy or during treatment with hormonal agents (i.e., luteinizing hormone-releasing hormone [LHRH] agonists)
* Elevated prostate-specific antigen (PSA) > 2 ng/mL and PSA progression after at least 12 weeks treatment with docetaxel/prednisone, within 90 days after discontinuation of docetaxel/prednisone treatment, under continued hormonal treatment (i.e., LHRH agonists or orchiectomy), and meets 1 of the following criteria for PSA progression:

  * PSA increase of ≥ 25% above the nadir
  * PSA increase of ≥ 25% above the baseline if no decrease has been observed

    * The increase is a minimum of 2 ng/mL, and it is confirmed 1 week later
* No presence or history of CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Neutrophils ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN
* Creatinine clearance ≥ 30 mL/min
* Patient compliance and geographic proximity allow proper staging and follow-up
* Peripheral neuropathy < grade 2
* No prior malignancy within the past 5 years with the exception of localized nonmelanoma skin cancer or Ta or Tis bladder cancer
* No known hypersensitivity to trial drugs or any of their components
* No serious underlying medical condition that, in the judgment of the investigator, would preclude the patient's ability to participate in the trial (e.g., active autoimmune disease, uncontrolled or acute severe infection, or uncontrolled diabetes)
* No psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, or interfering with oral drug intake compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior radiotherapy
* More than 6 weeks since prior treatment with antiandrogens (i.e., flutamide or bicalutamide)
* No prior chemotherapy other than docetaxel for metastatic prostate cancer
* No other concurrent experimental drugs or other anticancer therapy

  * Concurrent bisphosphonates and LHRH agonists allowed provided these medications started at least 2 months prior to study therapy
* No treatment in a clinical trial within the past 30 days
* No prior treatment with drugs interacting with epidermal growth factor receptor (i.e., cetuximab, panitumumab, gefitinib, erlotinib hydrochloride, or multi-tyrosine kinase inhibitors)
* No concurrent drugs that, according to the Swissmedic-approved product information, are contraindicated for use with the trial drugs

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | at 12 weeks
Progression-free survival (PFS) | at 24 weeks

SECONDARY OUTCOMES:
Adverse events | All AEs will be assessed according to NCI CTCAE v3.0.
Prostate-specific antigen (PSA) response (30% and 50% PSA response) | is defined as a decrease in PSA level of at least 50% (compared to baseline PSA) confirmed after 3-4 weeks (according to the PSA working group consensus criteria)
Tumor assessment of measurable disease according to RECIST criteria | after 12 weeks of treatment, or earlier if clinically indicated
Tumor assessment of bone lesions | at 12 weeks
Overall survival | calculated from registration until death.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cathomas, MD, Study Chair — Kantonsspital Graubuenden; Roger von Moos, MD, Principal Investigator — Kantonsspital Graubuenden; Silke Gillessen, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (21):
- Switzerland (21):
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Bruderholz, Bruderholz
  - AndreasKlinik Cham Zug, Cham
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Freiburg, Fribourg
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital, Luzerne, Luzerne
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum, Zurich
  - Klinik Hirslanden, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Cathomas R, Rothermundt C, von Moos R, et al.: Cetuximab in combination with docetaxel in patients (pts) with metastatic castration resistant (mCRPC) and docetaxel-refractory prostate cancer: A multicenter phase II trial (SAKK 08/07). [Abstract] J Clin Oncol 28 (Suppl 15): A-4666 , 2010.
- [Result] Cathomas R, Rothermundt C, Klingbiel D, Bubendorf L, Jaggi R, Betticher DC, Brauchli P, Cotting D, Droege C, Winterhalder R, Siciliano D, Berthold DR, Pless M, Schiess R, von Moos R, Gillessen S; Swiss Group for Clinical Cancer Research SAKK. Efficacy of cetuximab in metastatic castration-resistant prostate cancer might depend on EGFR and PTEN expression: results from a phase II trial (SAKK 08/07). Clin Cancer Res. 2012 Nov 1;18(21):6049-57. doi: 10.1158/1078-0432.CCR-12-2219. Epub 2012 Sep 12. PMID 22977195